CLINICAL TRIAL: NCT05715398
Title: A Multicenter, Open Phase Ⅰ/Ⅱa Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of BR790 in Combination With Anlotinib in Subjects With Advanced Non-small Cell Lung Cancer
Brief Title: BR790 in Combination With Anlotinib in Adult Subjects With Advanced Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Gopherwood Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR790-103
Record Dates: First submitted 2023-01-12; First posted 2023-02-08 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: BR790; Anlotinib; NSCLC; PTPN11; SHP2
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Noonan Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BR790+anlotinib (Experimental): BR790 will be administered orally, variable dose on Day 1 of each 21-day cycle, Anlotinib will be administered as PO fixed dose on Day1-14 of each 21-day cycle
  Interventions: Drug: BR790+anlotinib

INTERVENTIONS:
Drug: BR790+anlotinib — BR790 will be administered orally, variable dose on Day 1 of each 21-day cycle， Anlotinib will be administered as PO fixed dose on Day1-14 of each 21-day cycle

SUMMARY:
This is a Phase Ⅰ/Ⅱa, multi-center, open-label study, aiming to evaluate the safety, tolerability, pharmacokinetic (PK), and efficacy of BR790 in combination with anlotinib in adult participants with advanced NSCLC.

DETAILED DESCRIPTION:
This study is a Phase Ⅰ/Ⅱa, multi-center, open-label study of BR790 in combination with anlotinib with a dose escalation part followed by a dose expansion part in adult subjects with advanced NSCLC. Participants will be treated until disease progression per RECIST v1.1, unacceptable toxicity, or other criteria for withdrawal are met, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤75 years old.
* Subjects with histologically or cytologically confirmed locally advanced or relapsed metastatic driver negative (EGFR, ALK, ROS, etc.) advanced NSCLC，whose disease progressed after at least 2 previous standard therapies.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Has at least one measurable lesion per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) .

Exclusion Criteria:

* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has uncontrolled moderate to massive effusion.
* Central lung squamous carcinoma along with cavum, or non-small cell lung cancer along with hemoptysis (>50ml/day).
* Other kinds of malignancies within 5 years or for now.
* Has not enough organ functional reserve at baseline, which met at least one of the following criteria： ANC<1.5×10^9/L, PLT<100×10^9/L, Hb<100g/L; TBIL>1.5×ULN, ALT or AST>2.5×ULN (without liver metastases) , ALT or AST>5×ULN (with liver metastases);Cr >1.5×ULN, urine protein≥++，or confirmed 24h urine protein≥1.0g;INR >1.5×ULN, PT>1.5ULN or APTT >1.5×ULN.
* Previous use of other SHP2 inhibitors (such as TNO-155, JAB-3312, JAB-3068, RLY-1971, RMC-4630, etc.)
* Has used anlotinib before
* The first assessment of efficacy was PD, or occurred ≥grade 3 adverse reactions with antitumor angiogenesis small-molecule drugs (e.g. Apatinib, surufatinib, fruquintinib, etc.), or less than 6 months after the last antitumor vascular therapy.
* Has got non remissive toxic reactions derived from previous therapies, which is over level 1 in CTC AE (5.0), alopecia and grade 2 peripheral neuropathy are not included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose/Recommended Phase Ⅱ Dose(MTD/RP2D) | 2 years
  To evaluate the MTD/RP2D of BR790 in combination with anlotinib (Part 1)
Objective Response Rate (ORR) | 2 years
  To evaluate the objective response rate (ORR) of BR790 in combination with anlotinib. ORR is defined as the proportion of subjects who achieve a Complete Response (CR) or Partial Response (PR) as assessed by RECIST v1.1 (Part 2)

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years
  PFS was defined as the time from randomization to documented disease progression per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) or death due to any cause, whichever occurred first.
Duration of overall response (DOR) | 2 years
  DOR is defined as the time from the first documented CR or PR per RECIST v1.1 to disease recurrence or disease progression (PD) whichever occurs first.
Disease Control Rate(DCR) | 2 years
  DCR is defined as the proportion of subjects who achieve a Complete Response (CR) 、Partial Response (PR) or Stable Disease (SD) as assessed by RECIST v1.1
Overall Survival (OS) | 2 years
  OS is defined as the time from study treatment initiation to death from any cause or last day known to be alive.
Adverse Events(AEs) | 2 years
  Incidence, nature, and severity of treatment-emergent AEs and serious AEs, including incidence and severity of findings in laboratory values and vital signs for combination therapy
Area under the plasma concentration-time curve (AUC) | 2 years
  Area under the plasma concentration time curve of BR790/anlotinib
Plasma concentration (Cmax) | 2 years
  Highest observed plasma concentration of BR790/anlotinib

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, Principal Investigator — Shanghai Chest Hospital

IPD SHARING:
Plan to Share IPD: No